CLINICAL TRIAL: NCT03347630
Title: Prospective Evaluation of MRI in Pre-operative Staging of Esophagus Cancers
Brief Title: Pre-operative MRI of Esophagus Cancer
Acronym: STIRMCO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dromain Clarisse (Other)
Responsible Party: Sponsor-Investigator, Dromain Clarisse, MD, phD, University of Lausanne Hospitals
Organization: University of Lausanne Hospitals (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CER-VD 2017-00388; 17_015 (Other: CRC CHUV)
Record Dates: First submitted 2017-11-15; First posted 2017-11-20 (Actual); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Esophagus Cancer; Diagnoses Disease
Keywords: MRI; oesophagus cancer; Staging
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- oesophagus cancer MRI (Other): Diagnostic test
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — Thoraco-abominal MRI

SUMMARY:
The role of MRI in the management of esophageal cancer remains unclear and poorly studied. Recent technical advances suggest that MRI may become a powerful technique for the initial assessment of esophageal cancer, but also for the evaluation of response to neo-adjuvant treatment before surgery.

This imaging study will be performed prospectively and consecutively in 60 patients included over a 18-month period in patients wîth newly diagnosed esophageal cancer.

The aim of this study is to assess the accuracy of MRI to visualize esophageal tumors, to assess tumor burden and potential contact with adjacent structures as well as associated lymph nodes. If chemotherapy or radio-chemotherapy treatment is indicated before surgery, we will also evaluate whether MRI helps us to better evaluate the response to this treatment in comparison to PET-scan or echo. endoscopy which are the examinations currently performed to evaluate the effectiveness of these treatments.

The images of the MRI exams will be interpreted by 1 expert radiologist with no knowledge of the other imaging modalities and transmitted to the doctors in charge for possible consideration for the treatment.

Patients will then be followed for one year according to clinical management standards to study the data on treatment complications and cancer progression at one year.

The main risk is the administration of a gadolinium chelate-based MRI contrast product used routinely. There is also a risk that the results of the MRI may influence the treatment initially planned for example by canceling a surgical procedure.

DETAILED DESCRIPTION:
The study will be proppsed consecutively to all patients with a histologically proven diagnosis of esophageal cancer.

An MRI examination including morphological sequences (without and with injection of a gadolinium chelate) functional and dynamic will be carried out in all the patients for initial staging in addition to other diagnostic procedure performed in clinical routine in this indication that are the endo-ultrasonography, CT and PET scanner.

In patients for whom neo-adjuvant treatment with chemotherapy or radio-chemotherapy will be decided and started, a second MRI will be performed 4 to 6 weeks after the end of the neo-adjuvant treatment.

The images of the MR exams will be interpreted by 1 expert radiologist blinded from data of other imaging modalities and transmitted to the doctors in charge of the patient for possible consideration for the treatment.

Patients will then be followed for one year according to regular recommandation to assess mortality / morbidity and PFS at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Any pathologically proven oesophagus cancer

Exclusion Criteria:

* MRI contraindication
* Pregnant women
* cervical esophagus cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-10-02 (Actual); Primary Completion 2018-10-01 (Estimated); Study Completion 2019-03-30 (Estimated)

PRIMARY OUTCOMES:
diagnostic performance for staging | 18 months
  TNM staging

SECONDARY OUTCOMES:
Diagnostic performance for staging | 18 months
  Assessment of rate of Under and overstaging
Prognostic biomarker | 18 months
  correlation of MRI data with PFS, morbidity mortality rate and surgical resection
Diagnostic performance to assess tumor response | 18 months
  Correlation of changes of ADC values and histological TRG

CONTACTS AND LOCATIONS:
Overall Officials: Clarisse Dromain, MD, phD, Principal Investigator — CHUV
Locations (1):
- CHUV, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No